CLINICAL TRIAL: NCT01613989
Title: Total Hip Prosthesis Assisted by Computer Based on Pre-operative EOS Imaging
Brief Title: Total Hip Prosthesis Assisted by Computer
Acronym: NAVEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2011/07
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Clinic Hip Osteoarthrosis
Keywords: Hip arthroplasty; navigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Active Comparator): Reference group, installation of hip prothesis following standard procedure
  Interventions: Procedure: Prosthetic hip surgery, operated under manual control
- Treatment 2 (Active Comparator): :treatment group,installation of hip prosthesis with assistance by computer based on imaging EOS
  Interventions: Procedure: Prosthetic hip surgery operated under navigation based on EOS imaging

INTERVENTIONS:
Procedure: Prosthetic hip surgery, operated under manual control — : Hip replacement is performed in supine side position. Cup is positioned under manual control with the aid of a manual ancillary.
  Arms: Treatment 1
Procedure: Prosthetic hip surgery operated under navigation based on EOS imaging — The patient will be installed in supine side position. The cup will be navigated with the technique based on EOS imaging. This technique requires the registration of the homolateral antero superior iliac spine and the homolateral postero superior iliac spine only. It does not require the registration of the pubis or any other controlateral points which are poorly accessible in the supine side position
  Arms: Treatment 2

SUMMARY:
Computer assistance in prosthetic hip surgery is able to improve the accuracy of the surgery: Associating hip navigation and EOSTM imaging pre-operatively could simplify the procedure of hip navigation in lateral decubitus while maintaining the accuracy of the technique

DETAILED DESCRIPTION:
Hip navigation based on preoperative EOS(TM) imaging could help to improve the accuracy of cup positioning like other computer assisted hip surgery, but it would also simplify the procedure in lateral decubitus. Indeed, the registration of the controlateral antero superior iliac spine and the pubis is not necessary with this technique. The target population of the study is the one affected with primitive hip osteoarthritis for which an indication of prosthesis of total hip has been chosen Expected Result: Simplification of the procedure of navigation of the cup. Decrease in the number of cups positioned out of the "security zone" compared to the standard manual technique of cup positioning. A result of 50% of good positioning is expected with the manual technique versus 80% with the technique of navigation based on EOS(TM).

MAIN OBJECTIVE: Compare the surgical treatment of total hip prosthesis without assistance by computer and total hip prosthesis with navigation based on imaging EOSTM pre-operative Comparative clinical trial of superiority, randomized in single blind, in 2 parallel groups: -Group 1: Installation of hip prosthesis without assistance by computer -Group 2: Installation of hip prosthesis with assistance by computer based on imaging EOS(TM)

ELIGIBILITY:
Inclusion Criteria:

* Nosologic criteria :
* Primitive clinic hip osteoarthrosis
* secondary secondary clinic hip osteoarthrosis : osteonecrosis of femoral head posttraumatic
* Primitive radiological hip osteoarthrosis,
* Indication of total hip prosthesis
* Free informed and written consent, dated and signed by the patient and the investigator before any examination required by the research
* Subject affiliated or beneficiary of the social security
* Man or woman aged from 40 to 90 years

Exclusion Criteria:

* The navigation based on EOSTM imaging. requires the visualization on the EOSTM. pre-operative radiography of 6 radiological bone markers. The non-viewing of these markers is a criterion for exclusion of the study.
* anaesthetic contraindication
* pregnant women
* Persons under the control of justice

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2014-11-06 (Actual); Study Completion 2014-11-06 (Actual)

PRIMARY OUTCOMES:
Positioning of the cup in the 'security zone'. Comparison performed in immediate post-operative | The measure of the positioning of the cup will be carried out on the control scanner post-operatively at 3 months

SECONDARY OUTCOMES:
Post-operative dislocation | at 1 year of the occurrence of at least 1 episode of dislocation post-operatively
  propotion of Post-operative dislocation : Comparison at 1 year of the occurrence of at least 1 episode of dislocation post-operatively
Functional Score of Harris and the score PMA | at 3 month,6 month, and 12 months
  mean of Functional Score of Harris and the score PMA
Quality of live score | at 3 month,6 month,and 12 months
  . Quality of live score: Womac score, SF12,Oxford Score: comparison at 3 month,6 month,one year Measure : expressed as a mean
Early sign of radiographic unsealing | comparison at one year
  Early sign of radiographic unsealing : comparison at one year 2 blinded operators Measure : expressed as a mean
Average surgical Time | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Anselme BILLAUD, Principal Investigator — University Hospital Bordeaux, France; Anntoine BENARD, Study Chair — University Hospital Bordeaux, France
Locations (1):
- Unité d'orthopédie-traumatologie, membre supérieur CHU Pellegrin, Bordeaux, France